CLINICAL TRIAL: NCT07305129
Title: Pressure-Controlled Versus Volume-Controlled Ventilation in Low-Flow Anesthesia: A Randomized Controlled Trial on Intraoperative Respiratory Mechanics and Postoperative Pulmonary Function
Brief Title: PCV vs VCV in Low-Flow Anesthesia
Status: Completed | Type: Observational
Sponsor: HULYA TOPCU, MD (Other)
Responsible Party: Sponsor-Investigator, HULYA TOPCU, MD, Assoc. Prof. MD, Erol Olcok Corum Training and Research Hospital
Organization: Erol Olcok Corum Training and Research Hospital (Other)
Other Study IDs: 2023-64; hulya topcu (Other: Erol Olcok Corum Training and Research Hospital); serhat ozciftci (Other: Erol Olcok Corum Training and Research Hospital)
Record Dates: First submitted 2025-11-27; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-10

CONDITIONS: ASA Class I/II Patients; General Anesthetic; Low Flow Anesthesia
Keywords: low-flow anesthesia; pressure-controlled ventilation; volume-controlled ventilation; respiratory mechanics; peak inspiratory pressure; pulmonary function

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this observational study is to investigate the effects of ventilation modes on intraoperative and postoperative lung functions in patients under general anesthesia.

This study aimed to compare the effects of low-flow anesthesia on intraoperative respiratory mechanics and early postoperative pulmonary function between PCV and VCV in ASA I-II adult patients.

DETAILED DESCRIPTION:
Studies comparing the effects of pressure-controlled ventilation (PCV) and volume-controlled ventilation (VCV) on lung function under low-flow conditions are limited. In this study, the effects of PCV and VCV on intraoperative respiratory mechanics and early postoperative pulmonary function were investigated during low-flow anesthesia in ASA I-II adult patients undergoing routine anesthesia procedures.

ELIGIBILITY:
Inclusion Criteria:

- age 18-65 years and American Society of Anesthesiologists (ASA) physical status I-II.

Exclusion Criteria:

* morbid obesity (BMI > 35 kg/m²),
* scoliosis or thoracic deformity,
* restrictive or obstructive lung disease,
* prior thoracic or upper abdominal surgery,
* history of major thoracic trauma or congenital chest wall anomaly,
* active smoking or chronic use of corticosteroids,
* β-agonists, bronchodilators, or antihistamines,
* anticipated difficult airway
* severe hypoxemia (SpO₂ < 90%) during induction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hitit University Erol Olçok Training and Research Hospital
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Mean Ppeak (cmH₂O) at each time point; between-group difference. | From post-intubation baseline until 30 minutes after initiation of low-flow anesthesia (approximately 45 minutes total).
  Peak inspiratory pressure will be measured using the anesthesia workstation's built-in pressure monitoring system. Ppeak (cmH₂O) values will be automatically recorded at predefined time points: baseline after intubation, before low-flow transition, and 5, 10, 15, and 30 minutes after transition to low-flow anesthesia. Group comparisons will be reported as mean ± SD and analyzed for intergroup differences.

SECONDARY OUTCOMES:
Change in inspiratory score (number of balls raised). | Baseline to 30 minutes after initiation of low-flow anesthesia and Preoperative baseline and postoperative 1 hour
  Mean airway pressure will be measured continuously by the anesthesia machine. Values will be recorded at the same predefined time points as Ppeak. Data will be reported as mean ± SD. Dynamic compliance (mL/cmH₂O) will be calculated using the ventilator's automated measurement system (tidal volume / (Ppeak - PEEP)). Values will be recorded at identical intraoperative time points. Data will be reported as mean ± SD. Inspiratory effort will be assessed using the Triflo incentive spirometer by recording the number of balls elevated on a single maximal inspiratory attempt (range: 0-3). Measurements will be taken preoperatively and 1 hour postoperatively in the recovery unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Hitit University Erol Olçok Training and Research Hospital, Çorum, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided